CLINICAL TRIAL: NCT02626793
Title: Long-term Documentation of the Utilization of Otezla® in Patients With Plaque Psoriasis Under Routine Conditions (LAPIS-Pso)
Brief Title: A Study of Otezla® in Patients With Plaque Psoriasis Under Routine Conditions
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: CC-10004-PPSO-002
Record Dates: First submitted 2015-07-29; First posted 2015-12-10 (Estimated); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Psoriasis
Keywords: Plaque psoriasis; Apremilast; Otezla®; LAPIS-Pso; Observational; CC-10004; non-interventional; Germany
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with ≤ 1 conventional, systemic pre-treatment: After failure (inadequate response/intolerance) to or contraindication for ≤ 1 conventional, systemic pre-treatment
- Patients with > 1 conventional, systemic pre-treatment: After failure (inadequate response/intolerance) to or contraindication for > 1 conventional, systemic pre-treatment

SUMMARY:
The objective of this NIS is the collection of data on the utilization of Apremilast under routine conditions in Germany. Patients' quality-of-life and treatment satisfaction on treatment with Apremilast in daily practice will be documented. Moreover, physician's and patient's assessments of the effectiveness and safety of Apremilast will be recorded. FPI was 3rd August 2015, LPO was 14th of June 2018. A total of 391 patients have been enrolled.

DETAILED DESCRIPTION:
The objective of this NIS (according to section 4(23) of the German Medicinal Products Act) is the documentation of data on the effectiveness and tolerability of an Apremilast treatment under routine clinical conditions in German patients with plaque psoriasis.

This NIS is intended to reflect the apremilast treatment of patients with plaque psoriasis who have received at least one prior conventional, systemic therapy or, if a contraindication is present, did not receive a systemic therapy so far, and who were diagnosed by their treating physicians to be eligible for an apremilast treatment. The treatment of Apremilast will be documented for a period of approximately 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* The decision for a therapy with Apremilast was made before enrolment and independent of this study.
* Patient ≥ 18 years of age
* Diagnosis of moderate to severe plaque psoriasis
* Inadequate response or intolerance to a previous systemic treatment, or contraindication for systemic therapies.
* Written informed consent by the patient for data recording, statistical analysis, filing and forwarding of the data

Exclusion Criteria:

* Pregnancy
* Hypersensitivity to apremilast or any of the excipients of the film-coated tablet
* Other criteria according to the Summary of product characteristics (SmPC).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 500 patients with moderate to severe plaque psoriasis are planned to be enrolled in this NIS. In- and exclusion criteria are derived from the Summary of product characteristics (SmPC) of Apremilast.
Sampling Method: Non-Probability Sample
Enrollment: 391 (Actual)
Dates: Start 2015-08-03 (Actual); Primary Completion 2017-06-08 (Actual); Study Completion 2018-06-14 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the Dermatology Life Quality Index (DLQI) ≤ 5 or improvement in DLQI by ≥ 5 points at Visit 2 from baseline | Approximately 4 months
  DLQI is a simple, compact, and practical questionnaire for use in a dermatology clinical setting to assess limitations related to the impact of skin disease. The instrument contains ten items dealing with the participant's skin. With the exception of Item Number 7, the participant responds on a four-point scale, ranging from "Very Much" (score 3) to "Not at All" or "Not relevant" (score 0). Item Number 7 is a multi-part item, the first part of which ascertains whether the participant's skin prevented them from working or studying (Yes or No, scores 3 or 0 respectively), and if "No," then the participant is asked how much of a problem the skin has been at work or study over the past week, with response alternatives being "A lot," "A little," or "Not at all" (scores 2, 1, or 0 respectively). The DLQI total score is derived by summing all item scores, which has a possible range of 0 to 30, with 30 corresponding to the worst quality of life, and 0 corresponding to the best.

SECONDARY OUTCOMES:
Change from Baseline in the Dermatology Life Quality Index (DLQI) ≤ 5 or improvement in DLQI by ≥ 5 points at all other visits from baseline. | Up to approximately 52 weeks
  DLQI is a simple, compact, and practical questionnaire for use in a dermatology clinical setting to assess limitations related to the impact of skin disease. The instrument contains ten items dealing with the participant's skin. With the exception of Item Number 7, the participant responds on a four-point scale, ranging from "Very Much" (score 3) to "Not at All" or "Not relevant" (score 0). Item Number 7 is a multi-part item, the first part of which ascertains whether the participant's skin prevented them from working or studying (Yes or No, scores 3 or 0 respectively), and if "No," then the participant is asked how much of a problem the skin has been at work or study over the past week, with response alternatives being "A lot," "A little," or "Not at all" (scores 2, 1, or 0 respectively). The DLQI total score is derived by summing all item scores, which has a possible range of 0 to 30, with 30 corresponding to the worst quality of life, and 0 corresponding to the best.
Change in the Physician Global Assessment (PGA) Score | Up to approximately 52 weeks
  The PGA is a 5-point scale ranging from 0 (clear), 1 (almost clear), 2 (mild), 3 (moderate), to 4 (severe), incorporating an assessment of the severity of the Plaque-Psoriasis.
Percent Change in Percent of Affected Body Surface Area (BSA) | Up to approximately 52 weeks
  BSA is a measurement of involved skin. The overall BSA affected by psoriasis is estimated based on the palm area of the participant's hand (entire palmer surface or "handprint" excluding DIPs), which equates to approximately 1% of total body surface area.
Percent Change in the Psoriasis Area Severity Index (PASI) Score | Up to approximately 52 weeks
  Psoriasis Area Severity Index (PASI) scores range from 0 to 72, with higher scores reflecting greater disease severity. Erythema, thickness, and scaling are scored on a scale of 0 (none) to 4 (very severe) on 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. Degree of involvement on each of the 4 anatomic regions is scored on a scale of 0 (no involvement) to 6 (90% to 100% involvement). The total qualitative score (sum of erythema, thickness, and scaling scores) is multiplied by the degree of involvement for each anatomic region and then multiplied by a constant. These values for each anatomic region are summed to yield the PASI score.
Change in the Patient's Global Assessment (PaGA) | Up to approximately 52 weeks
  The PaGA is a 5-point scale ranging from 0 (clear), 1 (almost clear), 2 (mild), 3 (moderate), to 4 (severe), incorporating an assessment of the severity of the Plaque-Psoriasis by the patient.
Patient Preference Questionnaire (PPQ) | Approximately 4 months
  PPQ is a questionnaire consisting of 5 questions. PPQ asks the patient for his preference of the actual therapy versus the previous systemic therapy.
Patient Satisfaction (Systemic Therapy Adherence Questionnaire, STAQ) | Approximately 13 months
  STAQ; patient questionnaire on patient benefit, communication physician/patient, patient knowledge, and treatment satisfaction with the current systemic treatment (38 questions).
Change in Pain (Visual Analogue Scale; VAS) | Up to approximately 52 weeks
  The Pain Visual Analog Scores (VAS) is used to measure the amount of pain a participant experiences. Participants are asked: How much pain do you actually experience? All VAS values range from 0 to 100. Higher scores correspond to more severe symptom or disease.
Adverse Events (AEs) | Up to approximately 52 weeks
  All Serious Adverse Events (SAEs), irrespective of relationship to Apremilast, and all non-serious AEs considered at least possibly related to Apremilast administration [non-serious adverse drug reactions (NS ADRs)], must be recorded within 24 hours of the physician's knowledge to the Sponsors' Drug Safety Department. AEs will be reported by the sponsor as required to Regulatory Authorities and Ethics Committees as applicable, in accordance with the national requirements for marketing authorization holders.
Change in Itch (Pruritus) (Visual Analogue Scale; VAS) | Up to approximately 52 weeks
  The Itch Visual Analog Scores (VAS) is used to measure the amount of itch a participant experiences. Participants are asked: How much itch do you actually experience? All VAS values range from 0 to 100. Higher scores correspond to more severe symptom or disease.
Change in Scalp Involvement -Physician's Global Assessment (PGA) | Up to approximately 52 weeks
  PGA: 5-point scale for the physician's global assessment of the severity of scalp psoriasis.
Change in Scalp Involvement - Patient's Global Assessment (PaGA) | Up to approximately 52 weeks
  PaGA: 5-point scale for the patient's global assessment of the severity of scalp psoriasis.
Change in Nail Involvement - Target Nail Psoriasis Severity Index (NAPSI) | Up to approximately 52 weeks
  NAPSI: Assessment of target fingernail for nail bed and nail matrix involvement, each can be scored 0-4. Total score ranges from 0-8.
Change in Nail Involvement Fingernail - Patient's Global Assessment (PaGA) | Up to approximately 52 weeks
  Fingernail Patient Global Assessment ; 5-point scale on the patient's global assessment of the fingernail involvement, substituted with a 0-100 Visual analog scale (VAS) for the assessment of the impairment caused by this nail involvement.
Change in Palmoplantar involvement - Palmoplantar physician's global assessment (PGA) | Up to approximately 52 weeks
  PGA: 5-point scale for the physician's global assessment of the severity of palmoplantar involvement.
Change in Palmoplantar involvement - Palmoplantar patient's global assessment (PaGA) | Up to approximately 52 weeks
  PaGA: 5-point scale for the patient's global assessment of the severity of palmoplantar involvement.

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (96):
- Germany (96):
  - Gertraud Krähn-Senftleben, Blaubeuren Abbey, Baden-Wurttemberg
  - Ralf-Uwe Peter, Blaustein, Baden-Wurttemberg
  - Regina Renner, Esslingen am Neckar, Baden-Wurttemberg
  - Universitätsklinikum Heidelberg - Hautklinik, Heidelberg, Baden-Wurttemberg
  - Ina Reitenbach-Blindt, Karlsruhe, Baden-Wurttemberg
  - Kaiserstraße 231-233, Karlsruhe, Baden-Wurttemberg
  - Naomi Gerhardus, Karlsruhe, Baden-Wurttemberg
  - Johannes Glutsch, Karlsruhe, Baden-Wurttemberg
  - Beate Schwarz, Langenau, Baden-Wurttemberg
  - Astrid Schmieder, Mannheim, Baden-Wurttemberg
  - Katharina Wroblewska, Spaichingen, Baden-Wurttemberg
  - Michael Sticherling, Erlangen, Bavaria
  - Hjalmar Kurzen, Freising, Bavaria
  - Claus Jung, Germering, Bavaria
  - Clarissa Allmacher, Hersbruck, Bavaria
  - Ildiko Sugar-Bunk, Krumbach, Bavaria
  - Sabine Anders, München, Bavaria
  - Hortensia Pfannenstiel, München, Bavaria
  - Technische Universität München - Kilian Eyerich, München, Bavaria
  - Universitätsklinikum Regensburg, Regensburg, Bavaria
  - Andreas Eggert, Würzburg, Bavaria
  - Lars Freitag, Falkensee, Brandenburg
  - Förster-Funke-Allee 104, Kleinmachnow, Brandenburg
  - Silke Thies, Schwedt, Brandenburg
  - Christoph Hartl, Eltville, Hesse
  - Universitätsklinikum Frankfurt, Klinik für Dermatologie, Venerologie und Allergologie, Frankfurt am Main, Hesse
  - Pia Freyschmidt-Paul, Schwalmstadt, Hesse
  - Jutta Ramaker-Brunke, Braunschweig, Lower Saxony
  - Andreas Kleinheinz, Buxtehude, Lower Saxony
  - Marco Averbeck, Cloppenburg, Lower Saxony
  - Florian Schenck, Hanover, Lower Saxony
  - Ulrike Stein, Hanover, Lower Saxony
  - Holger Petering, Hildesheim, Lower Saxony
  - Silke Reinecke, Holzminden, Lower Saxony
  - Reinhard Knöll, Lüneburg, Lower Saxony
  - Christian Kock, Vechta, Lower Saxony
  - Gesundheitszentrum Winsen, Winsen, Lower Saxony
  - Andreas Timmel, Bergen auf Rügen, Mecklenburg-Vorpommern
  - Raimund Paech, Neubrandenburg, Mecklenburg-Vorpommern
  - Theaterplatz 9, Aachen, North Rhine-Westphalia
  - Isaak Effendy, Bielefeld, North Rhine-Westphalia
  - Volker Riesopp, Duisburg, North Rhine-Westphalia
  - Bernhard Korge, Düren, North Rhine-Westphalia
  - Herderstr.71 b, Düsseldorf, North Rhine-Westphalia
  - Dechant-Deckers-Straße 5-7, Eschweiler, North Rhine-Westphalia
  - Universitätsklinikum Essen, Essen, North Rhine-Westphalia
  - Christina Huerkamp, Euskirchen, North Rhine-Westphalia
  - Sebastian Rotterdam, Gelsenkirchen-Feldmark, North Rhine-Westphalia
  - Jörg Brinkmann, Gladbeck, North Rhine-Westphalia
  - Hautartzpraxis, Kleve, North Rhine-Westphalia
  - Rudolf Stadler, Minden, North Rhine-Westphalia
  - Rolf Ostendorf, Mönchengladbach, North Rhine-Westphalia
  - Athanasios Tsianakas, Münster, North Rhine-Westphalia
  - Stefanie Montag, Rheinbach, North Rhine-Westphalia
  - Hautarztpraxis, Steinfeldstr. 5, Stolberg, North Rhine-Westphalia
  - Oliver Mainusch, Velbert, North Rhine-Westphalia
  - Kurt-Kräcker-Str. 47, Wesel, North Rhine-Westphalia
  - Magnus Bell, Andernach, Rhineland-Palatinate
  - Ulrich Blaese, Bendorf, Rhineland-Palatinate
  - Schloss Straße 17, Koblenz, Rhineland-Palatinate
  - Petra Staubach-Renz, Mainz, Rhineland-Palatinate
  - Dirk Maaßen, Maxdorf, Rhineland-Palatinate
  - Marktstr. 20, Neuwied, Rhineland-Palatinate
  - Praxis für Haut- und Geschlechtskrankheiten - Allergologie - Am Johannisborn, Prüm, Rhineland-Palatinate
  - Ralph von Kiedrowski, Selters, Rhineland-Palatinate
  - Mohammad Asefi, Simmern, Rhineland-Palatinate
  - Karolin Schneider, Chemnitz, Saxony
  - Beatrice Gerlach, Dresden, Saxony
  - Liane John, Dresden, Saxony
  - Mary-Krebs-Straße 1, Dresden, Saxony
  - Stefan Beissert, Dresden, Saxony
  - Bernhard-Göring-Str. 162, Leipzig, Saxony
  - Riebeckstraße 65, Leipzig, Saxony
  - Schweizergartenstr. 2a, Wurzen, Saxony
  - Puschkinstr. 110, Eilenburg, Saxony-Anhalt
  - Franckestr. 1, Magdeburg, Saxony-Anhalt
  - Jens Ulrich, Quedlinburg, Saxony-Anhalt
  - Gabriela Fiedler, Weißenfels, Saxony-Anhalt
  - Harald Brüning, Kiel, Schleswig-Holstein
  - Universitätsklinikum Schleswig-Holstein, Lübeck, Schleswig-Holstein
  - Christian Meewes, Neumünster, Schleswig-Holstein
  - Jens Thieme, Artern, Thuringia
  - Mario Pawlak, Heilbad Heiligenstadt, Thuringia
  - Raoul Hasert, Berlin
  - Klaus Spickermann, Berlin
  - Jens Olaf Mielcke, Berlin
  - Albert-Einstein-Str. 2, Berlin
  - Hautarztpraxis Zahn, Berlin
  - Maria Manasterski, Berlin
  - Martin Miehe, Berlin
  - Uwe Schwichtenberg, Bremen
  - Matthias Augustin, Hamburg
  - Kristian Reich, Hamburg
  - Christian Mensing, Hamburg
  - Johannes-R.-Becher-Straße 24, Königs Wusterhausen
  - Florian Kreuziger, Vilshofen

REFERENCES:
- [Derived] Reich K, Korge B, Magnolo N, Manasterski M, Schwichtenberg U, Staubach-Renz P, Kaiser S, Roemmler-Zehrer J, Gomez NN, Lorenz-Baath K. Quality-of-Life Outcomes, Effectiveness and Tolerability of Apremilast in Patients with Plaque Psoriasis and Routine German Dermatology Care: Results from LAPIS-PSO. Dermatol Ther (Heidelb). 2022 Jan;12(1):203-221. doi: 10.1007/s13555-021-00658-x. Epub 2021 Dec 15. PMID 34913153
- See also: Expanded Access for CC-10004 — https://clinicaltrials.gov/ct2/show/NCT02626793?term=CC-10004-PPSO-002&rank=1